CLINICAL TRIAL: NCT04710888
Title: Muco-bioadhesive Gel Containing Basil Extract (Ocimum Basilicum) in the Management of Recurrent Aphthous Stomatitis: A Randomized Clinical Study
Brief Title: Basil Extract (Ocimum Basilicum) in the Management of Recurrent Aphthous Stomatitis
Acronym: RCT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, malak mohamed shoukheba, associate prof., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3
Record Dates: First submitted 2021-01-08; First posted 2021-01-15 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Oral Ulcer
Keywords: Aphthous Stomatitis; basil extract; endocan marker
MeSH Terms: conditions — Oral Ulcer; Stomatitis, Aphthous | interventions — Anti-Inflammatory Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- basil extract mucoadhesive gel (Experimental): 10 patients treated with mucoadhesive gel containing 2% of basil extract 4 times per day (test group) for 20 min after every meal and before going to bed.
  Interventions: Drug: use of basil extract gel in treatment of aphthus ulcer
- mucoadhesive placebo gel (Placebo Comparator): 10 patients treated by mucoadhesive gel without drug which was used as placebo (contains tragacanth gum, alcohol, sodium benzoate, and distilled water) 4 times per day
  Interventions: Other: muco adhesive placebo gel
- healthy patients (Sham Comparator): 10 healthy patients will be selected to participate in the study to test the salivary level of endocan in the healthy individuals (negative control group)
  Interventions: Other: no treatment

INTERVENTIONS:
Drug: use of basil extract gel in treatment of aphthus ulcer — This study aimed to evaluate the efficacy of basil extract (Ocimum basilicum) in the treatment of aphthous ulcers
  Other Names: anti inflammatory and immunomodulation effect of basil extract
  Arms: basil extract mucoadhesive gel
Other: muco adhesive placebo gel — mucoadhesive gel without drug which was used as placebo (contains tragacanth gum, alcohol, sodium benzoate, and distilled water) 4 times per day
  Other Names: placebo gel
  Arms: mucoadhesive placebo gel
Other: no treatment — (i) had underlying systemic disease(s) or a history of immunologic disorder(s); (ii) were taking immunomodulatory agents or systemic nonsteroidal anti-inflammatory drugs < 1 month before study commencement; (iii) are smokers; (iv) are pregnant; (v) had a history of abusing drugs or alcohol; (vi) could not provide written informed consent.
  Other Names: negative control
  Arms: healthy patients

SUMMARY:
A randomized double-blind placebo controlled trial will be carried out on 20 patients complaining from aphthus ulcer and 10 patient healthy control 10 patients treated with mucoadhesive gel containing 2% of basil extract 4 times per day (test group) for 20 min after every meal and before going to bed. The other 10 patients treated by mucoadhesive gel without drug which was used as placebo (composed from 6% w/w PVA (Mw = 31-50 kDa, 98-99% hydrolysed) and 2% w/w sodium tetraydroxy borate) 4 times per day 10 healthy patients will be selected to participate in the study to test the salivary level of endocan in the healthy individuals (negative control group)

DETAILED DESCRIPTION:
A randomized double-blind placebo controlled trial will be carried out on 20 patients complaining from aphthus ulcer and 10 patient healthy control. Inclusion criteria will be: (i) age > 18 years; (ii) a clear history of RAS(recurrent apthous stomatitis)occurring no less than four times a year; (iii) presentation with one or two ulcers measuring 10 mm in diameter for 48 hours and yet to receive treatment; (iv) ulcers that took > 5 days to resolve without treatment. Individuals will excluded if they: (i) had underlying systemic disease(s) or a history of immunologic disorder(s); (ii) were taking immunomodulatory agents or systemic nonsteroidal anti-inflammatory drugs < 1 month before study commencement; (iii) are smokers; (iv) are pregnant; (v) had a history of abusing drugs or alcohol; (vi) could not provide written informed consent.

10 patients treated with mucoadhesive gel containing 2% of basil extract 4 times per day (test group) for 20 min after every meal and before going to bed. The other 10 patients treated by mucoadhesive gel without drug which was used as placebo (composed from 6% w/w PVA (Mw = 31-50 kDa, 98-99% hydrolysed) and 2% w/w sodium tetraydroxy borate) 4 times per day 10 healthy patients will be selected to participate in the study to test the salivary level of endocan in the healthy individuals (negative control group)

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years;
* a clear history of RAS (recurrent apthous stomatitis) occurring no less than four times a year;
* presentation with one or two ulcers measuring 10 mm in diameter for 48 hours and yet to receive treatment;
* ulcers that took > 5 days to resolve without treatment.

Exclusion Criteria:

* had underlying systemic disease(s) or a history of immunologic disorder(s);
* were taking immunomodulatory agents or systemic nonsteroidal anti-inflammatory drugs < 1 month before study commencement;
* are smokers;
* are pregnant;
* had a history of abusing drugs or alcohol;
* could not provide written informed consent

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
pain score VAS (Visual Analogue Scale) | one week
  The patients will be asked to record the daily level of pain severity of the ulcers through VAS (Visual Analogue Scale). It consisted of a 10-cm horizontal line, and the end of the line is (0) indicating "no pain" and the other end is (10) denoting "unbearable pain".
healing duration | one week
  patient evaluated by how long the ulcer takes to heal from baseline
size of the ulcer | one week
  measuring the ulcer size at baseline,5 days, and one week
salivary endocan level | one week
  enzyme-linked immunosorbent assays to measure the salivary concentrations of endocan marker at the first visit (i.e., before treatment) and the other was just after healing

CONTACTS AND LOCATIONS:
Overall Officials: malak YM shoukheba, Principal Investigator — faculty of dentistry tanta university
Locations (1):
- Malak Yousef Mohamed Shoukheba, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes